CLINICAL TRIAL: NCT01257685
Title: Selenoprotein P and Non-alcoholic Fatty Liver Disease
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, Kyung Mook Choi, Professor, Korea University
Other Study IDs: SEPP1(NAFLD)
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Non-alcoholic Fatty Liver Disease; Insulin Resistance
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood samples. Abdominal VFA and total abdominal fat area were measured via CT scan without an intravenous contrast agent
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control Group: Normal group
- NAFLD Group: NAFLD in the present study was defined a value of LAI <5 HU using an unenhaned CT.

SUMMARY:
The pathogenesis of nonalcoholic fatty liver disease has not been fully elucidated. The most widely supported theory implicates insulin resistance as the key mechanism leading to hepatic steatosis, and perhaps also to steatohepatitis.

Selenoprotein P(SeP) is a secretory protein primarily produced by the liver. Previous studies demonstrated that SeP, a liver-derived secretory protein, causes insulin resistance.

Therefore, the purpose of this study is to determine the different Sep levels between healthy normal group and NAFLD group.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD), a disease spectrum that includes simple steatosis, nonalcoholic steatohepatitis (NASH) and cirrhosis, has been increasingly recognized as the hepatic manifestation of metabolic syndrome. Both inflammation and insulin resistance are considered to be pivotal pathogenic mechanisms of NAFLD, as well as metabolic syndrome, type 2 diabetes, and atherosclerosis. There is mounting evidence implicating adipokines secreted from adipose tissue in the pathogenesis and progression of NAFLD, in addition to the development of insulin resistance and inflammation. Selenoprotein P (SeP) has recently been reported as a novel hepatokine that regulates insulin resistance and systemic energy metabolism in rodents and humans. Although previous studies have shown a close relationship among insulin resistance, inflammation, and NAFLD, as far as we know, there is no previous report evaluating the association between SeP and NAFLD. In the present study, we examined serum SeP levels in subjects with increased visceral fat area (VFA) or liver fat accumulation measured with computed tomography (CT). We evaluated the relationship between SeP levels and cardiometabolic risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers for visiting routine medical check in our clinic

Exclusion Criteria:

* History of cardiovascular disease(myocardial infarction, unstable angina, or cardiovascular revascularization)
* Diabetes
* Hypertension
* Malignancy
* Severe renal or hepatic disease
* Subjects taking medications that might affect body weight or body composition

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers for visiting routine medical check in our clinic
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2007-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Association between SeP and NAFLD | through study completion, an average of 2 year
  We used multiple logistic regression analysis

SECONDARY OUTCOMES:
Compare SeP level between control and NAFLD group | through study completion, an average of 2 year
  using Mann-Whitney U test
Correlation between SeP level and cardiometabolic risk factors | through study completion, an average of 2 year
  SeP level was stratified by tertile.

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Mook Choi, MD.PhD, Study Director — Korea University
Locations (1):
- Hae Yoon Choi, Seoul, South Korea